CLINICAL TRIAL: NCT01099891
Title: The Clinical Study for Evaluation of Efficacy and Safety of EGF on Oral Mucositis in Radiation Therapy Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sang-wook, Lee, Asan medical center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_EGF010P
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Stomatitis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- EGF (Experimental)
  Interventions: Drug: rhEGF
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhEGF — rhEGF 50 μg/ml, spray type, twice a day
  Arms: EGF
Drug: Placebo — Placebo, Spray type, Twice a day
  Arms: Placebo

SUMMARY:
The purpose of this Study is to evaluate the efficacy and safety of rhEGF on oral mucositis in patients receiving the radiation therapy or the concurrent chemo-radiotherapy

DETAILED DESCRIPTION:
Radiation therapy causes many side effects especially oral mucositis. The purpose of this Study is to evaluate the efficacy and safety of rhEGF on oral mucositis in patients receiving the radiation therapy or the concurrent chemo-radiotherapy. Head and neck cancer patients who have a plan to receive a minimum of 50 Gy radiation therapy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy during the study period or females of childbearing potential
* Have oral mucositis or other oral conditions at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe oral mucositis (RTOG garde 3 or 4) | 5 weeks(at the point of receiving 50 Gy radiation)

SECONDARY OUTCOMES:
Incidence and duration of ≥ grade 2, 3 (RTOG scale) oral mucositis | 5 weeks(at the point of receiving 50 Gy radiation)
Incidence and duration of ≥ grade 2, 3 (WHO scale) oral mucositis | 5 weeks(at the point of receiving 50 Gy radiation)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan medical center, Seoul
  - Seoul National Colleage & Hospital, Seoul